CLINICAL TRIAL: NCT00658593
Title: A Phase III Study of Gemcitabine Plus Capecitabine (GEMCAP) Versus Gemcitabine Alone in Advanced Biliary Cancer
Brief Title: Gemcitabine With/Out Capecitabine in Locally Advanced, Unresectable, or Metastatic Biliary Cancer
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: due to poor accrual
Sponsor: NCIC Clinical Trials Group (Network)
Responsible Party: Sponsor
Organization: Canadian Cancer Trials Group (Network)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BI1; CAN-NCIC-BI1 (Other: PDQ); CDR0000592854 (Other: PDQ)
Record Dates: First submitted 2008-04-12; First posted 2008-04-15 (Estimated); Last update posted 2023-08-04 (Actual); Status verified 2020-04

CONDITIONS: Extrahepatic Bile Duct Cancer; Gallbladder Cancer; Liver Cancer
Keywords: adenocarcinoma of the extrahepatic bile duct; unresectable extrahepatic bile duct cancer; recurrent extrahepatic bile duct cancer; adenocarcinoma of the gallbladder; adenocarcinoma with squamous metaplasia of the gallbladder; unresectable gallbladder cancer; recurrent gallbladder cancer; liver and intrahepatic biliary tract cancer
MeSH Terms: conditions — Bile Duct Neoplasms; Gallbladder Neoplasms; Liver Neoplasms; Carcinoma, Hepatocellular | interventions — Capecitabine; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GEMCAP (Active Comparator): Gemcitabine 1000mg/m2 IV days 1 and 8 ever 21 days; Capecitabine 650mg/m2 PO BID days 1-14 every 21 days.
  Interventions: Drug: capecitabine; Drug: gemcitabine hydrochloride; Procedure: quality-of-life assessment
- Gemcitabine Alone (Active Comparator): Gemcitabine 1000mg/m2 IV days 1, 8 and 15 every 28 days
  Interventions: Drug: gemcitabine hydrochloride; Procedure: quality-of-life assessment

INTERVENTIONS:
Drug: capecitabine
  Arms: GEMCAP
Drug: gemcitabine hydrochloride
Procedure: quality-of-life assessment

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as gemcitabine and capecitabine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. It is not yet known whether gemcitabine is more effective when given together with or without capecitabine in treating patients with biliary cancer.

PURPOSE: This randomized phase III trial is studying giving gemcitabine together with capecitabine to see how well it works compared with giving gemcitabine alone in treating patients with locally advanced, unresectable, or metastatic biliary cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To compare overall survival (OS) rates in patients with locally advanced, unresectable or metastatic biliary tree cancer treated with combined gemcitabine hydrochloride and capecitabine vs. gemcitabine hydrochloride alone.

Secondary

* To compare progression-free survival (PFS) in this patient group.
* To compare response rates (complete response [CR] and partial response [PR]) in this patient group.
* To compare stable disease (SD) rates in this patient group.
* To compare rate of disease control (CR, PR and SD) in this patient group.
* To estimate and compare response duration in this patient group.
* To compare the effects of these treatments on measures of quality of life in this patient group using the EORTC QLQ-C30.
* To compare the nature, severity and frequency of toxicities between the two arms.

OUTLINE: This is a multicenter study. Patients are stratified according to tumour type (cholangiocarcinoma vs. gallbladder or biliary unknown), ECOG performance status (0-1 vs. 2), extent of disease (locally advanced vs. metastatic), and treatment center. Patients are randomized to 1 of 2 treatment arms.

* Arm I (Gemcitabine hydrochloride and capecitabine): Patients receive gemcitabine hydrochloride IV on days 1 and 8 and oral capecitabine twice daily on days 1-14. Treatment repeats every 21 days in the absence of disease progression or unacceptable toxicity.
* Arm II (Gemcitabine hydrochloride alone): Patients receive gemcitabine hydrochloride IV on days 1, 8, and 15. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.

Quality of life is assessed at 12 weeks after randomization and 4 weeks after completion of study treatment.

After completion of study treatment, patients are followed at 4 weeks and then every 12 weeks thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically proven adenocarcinoma of the biliary tree (intra- and extra-hepatic biliary ducts or gallbladder)
* Locally advanced, unresectable, or metastatic disease

  * Patients with pathologically confirmed metastatic adenocarcinoma consistent with biliary primary with clinical documentation of gallbladder or biliary tree involvement and no evidence of another primary adenocarcinoma are eligible
* Must have evidence of disease but measurable disease is not required

  * Chest x-ray and/or CT scan of the chest, CT scan or MRI of the abdomen, and other radiological examination to document all disease sites have been done within 28 days prior to randomization

    * No repeat scan needed if a negative scan was performed within 35 days prior to randomization
  * Patients who have only one site of disease located inside a previous radiotherapy field are eligible

    * Lesions within a previous radiotherapy field may be considered measurable if documented ≥ 20% increase in size
    * If the lesion size increase has not been documented since the completion of radiotherapy, and the lesion is still present (i.e. not CR), the lesion is considered evaluable for this trial
* Patients with biliary duct obstruction are eligible provided all of the following criteria are met:

  * Treatable, clinically relevant obstruction
  * Obstruction has been relieved by internal endoscopic drainage/stenting, palliative bypass surgery or percutaneous drainage prior to trial entry
* No ampullary carcinomas (i.e., arising from the ampulla of Vater)
* No central nervous system (CNS) metastases, including active, progressive brain or leptomeningeal metastases

  * Patients with focal neurological symptoms must have had a CT scan to rule out CNS metastases

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Minimum life expectancy of 12 weeks
* Able (i.e. sufficiently fluent) and willing to complete the quality of life questionnaires in one of the validated languages
* Must be able to swallow and retain oral medication
* Hemoglobin > 90 g/L
* Absolute neutrophil count ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Total bilirubin < 3 times upper limit of normal(ULN)
* AST and/or ALT ≤ 5 times ULN
* Liver function tests stable and < 3 times ULN
* Serum creatinine < 160 µmol/L OR creatinine clearance > 60 mL/min
* Negative pregnancy test
* Fertile patients and their partners must agree to use adequate contraception prior to study entry, throughout the study, and for a period of 4 weeks after cessation of protocol therapy
* Patients must be accessible for treatment and follow-up
* No known dihydropyrimidine dehydrogenase deficiency
* No known hypersensitivity to gemcitabine or capecitabine
* No other active medical condition which would render the protocol treatment dangerous or impair the ability of the patient to receive protocol therapy, including, but not limited to, any of the following:

  * Unstable angina
  * Uncontrolled arrhythmia
  * Heart failure
* No other condition (e.g. psychological, geographical, etc.) that does not permit compliance with the protocol
* No other malignancies except adequately treated nonmelanoma skin cancer, curatively treated in-situ cancer of the cervix, or other solid tumors curatively treated with no evidence of disease for > 5 years

PRIOR CONCURRENT THERAPY:

* No prior chemotherapy for advanced or metastatic disease unless used in the following circumstances:

  * Fluorouracil or gemcitabine given concurrently with radiotherapy as a radiosensitizer, completed more than 3 months prior to randomization
  * Fluorouracil given as adjuvant treatment following surgery, completed at least 1 year prior to randomization
* No major surgery within 4 weeks of randomization
* No prior treatment with another investigational agent within 2 weeks of randomization
* At least 4 weeks from randomization since completion of prior radiotherapy and recovered

  * Patients may be randomized within the required 4 weeks if short course (< 5 fractions) of non-myelosuppressive radiotherapy was given
* Concurrent palliative radiation to a known site of bone metastasis allowed provided that the criteria for disease progression are otherwise not met
* No other concurrent anti-cancer therapy (cytotoxic, biological/immunotherapy or radiotherapy other than for known bone metastases as specified above)
* No other concurrent investigational drug therapy

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2008-10-10 (Actual); Primary Completion 2010-05-11 (Actual); Study Completion 2011-01-18 (Actual)

PRIMARY OUTCOMES:
Overall survival

SECONDARY OUTCOMES:
Progression-free survival
Response rates (complete response [CR] and partial response [PR])
Rate of stable disease (SD)
Rate of disease control (CR, PR, and SD)
Response duration
Quality of Life
Toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Knox, MD, Study Chair — Princess Margaret Hospital, Canada
Locations (8):
- Canada (8):
  - Tom Baker Cancer Centre - Calgary, Calgary, Alberta
  - Cross Cancer Institute at University of Alberta, Edmonton, Alberta
  - BCCA - Fraser Valley Cancer Centre, Surrey, British Columbia
  - British Columbia Cancer Agency - Vancouver Cancer Centre, Vancouver, British Columbia
  - Ottawa Hospital Regional Cancer Centre - General Campus, Ottawa, Ontario
  - St. Catharines General Hospital at Niagara Health System, St. Catharines, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - Hopital Charles Lemoyne, Greenfield Park, Quebec

IPD SHARING:
Plan to Share IPD: No